CLINICAL TRIAL: NCT03215901
Title: Life Plans of Young Adults in Rural KwaZulu-Natal: an Intervention Study
Brief Title: Life Plans Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Africa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-36591; 5K01MH105320 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-12 (Actual); Results first posted 2020-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2018-09

CONDITIONS: HIV/AIDS; Chronic HIV Infection; Health Knowledge, Attitudes, Practice
Keywords: Population-based survey; HIV treatment; HIV testing; Survival expectations; Condom use; Life plans; South African young adults
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A Beautiful Future Video (Experimental): Participants randomized to intervention will view intervention video.
  Interventions: Behavioral: A Beautiful Future Video
- Active Control Video (Sham Comparator): Participants randomized to control will watch a video of similar length as the intervention video on a different topic.
  Interventions: Behavioral: Active Control Video
- Pure Control (No Intervention): Participants view no video.

INTERVENTIONS:
Behavioral: A Beautiful Future Video — Video delivering information on the longevity gains due to HIV treatment in the area.
  Arms: A Beautiful Future Video
Behavioral: Active Control Video — Video on another topic.
  Arms: Active Control Video

SUMMARY:
The mass provision of HIV treatment in rural KwaZulu-Natal, South Africa has raised adult life expectancy by 18 years since 2003. We will conduct a population-based survey to assess young adults' beliefs about HIV, HIV treatment, and expectations for the future in the era of mass HIV treatment. Thh investigators will conduct a randomized evaluation to assess whether a short video providing young adults with information on longevity gains from HIV treatment affects young adults survival expectations, hope for the future, and health and educational behaviours, including uptake of HIV testing, the study's primary outcome.

DETAILED DESCRIPTION:
The proposed study will investigate survival expectations and health behaviours among young adults ages 18 to 25. Potential respondents will be sampled at random from a population listing from the demographic and health surveillance system of the Africa Health Research Institute (AHRI) in Somkhele, South Africa. Potential participants will be visited at home to be recruited for the study.

1. Consent. The study will be described and participants will provide written informed consent to participate in the study, including the baseline visit, a follow-up survey, and permission to link with demographic surveillance data.
2. Baseline interview (1.5 hours)

2.a) Survey module. First, a survey questionnaire will be conducted with young adults ages 18 to 25 to learn about their survival expectations, perceptions of HIV risks and treatment, future-oriented behaviours such as smoking, alcohol use, HIV risk behaviors, savings, locus of control, mental health, time and risk preference, and life satisfaction.

2.b) Video intervention. After the survey module, study participants will be randomized into treatment and control groups. Both interview participants and interviewers will be blinded to treatment assignment prior to this stage. The treatment group will be shown a 10 minute video that provides information on the changes in HIV-related mortality and life expectancy in the Demographic Surveillance Area between 2003 and today (an increase of about 18 years in the average length of life). The video includes testimonials from community members who have lived long and fulfilling lives on HIV treatment. The goal of the video is to increase measured survival expectations, hope, locus of control, and future orientation. The control group will receive a 10-minute video clip on another topic. Participants will be asked briefly for an open-ended response to the video: "what did the video make you think about?" which will be transcribed or recorded.

Details on randomization procedures: treatment assignment will be determined at the level of the household, such that if there are multiple respondents per household, they receive the same treatment. Households will be randomized to the intervention video or control ex ante. Though treatment assignment will occur ex ante, it will only be revealed - to both the field workers and the respondents - after completing the initial survey module. Ex ante randomization has two benefits. First, as a quality control, ex ante randomization limits the opportunity for violations of treatment assignment. Second, it increases power by enabling stratification on baseline variables. Because the study is nested in the AHRI population surveillance, treated and control households can be balanced on household size, wealth, and other characteristics. Treated and controls will be randomized at a 1:1 ratio, with controls further sub-randomized 1:1 to attention-placebo vs. pure control.

2.c) Re-survey module. Immediately after the video intervention, all study participants will be asked a brief subset of the survey module questions to re-measure survival expectations, locus of control, and life satisfaction. This step will estimate the immediate impact of the video intervention on beliefs.

2.d) Uptake of investment behaviors. 2.d.i) HIV Testing Voucher. Immediately after the re-survey module, participants will be offered a voucher for free HIV testing at a local pharmacy. Redeemed voucher numbers will be collected from the pharmacy to assess uptake of testing. No test results will be collected. This information will be stated clearly on the voucher.

2.d.ii) Invitation to Job Search Skills Workshop. Participants will be invited to a job skills training workshop delivered in partnership with a local human resources consultant. The workshop will inform participants of the types of job opportunities that exist, what skills and qualifications employers are looking for, as well as what strategies can be used to increase chances of getting a job. (For example, recent research in South Africa finds that employers are 60% more likely to respond to job applicants that include a letter of reference.) The workshop will be held at a convenient location 1-3 weeks after the baseline interview and attendance of study participants will be recorded. R10 will be provided to attendees to assist with travel expenses. The goal is to measure differences in uptake across treated and control arms, which will provide short-run evidence of the impact of the video on human capital investment behaviours.

2.d.iii) Savings choice. Immediately after the giving participants the HIV testing voucher, all participants will be offered the opportunity to save a portion of their participation compensation (R100) using a labelled box with a key that we will provide them. We provide this choice for study participants so that we can immediately measure intentions for future-oriented behaviour and to estimate the video's short-term effect based on differences in savings chosen between the treatment and control group.

2.d.iv) Condom offer. Participants will be offered the opportunity to purchase discount condoms and the number purchased will be recorded.

3. Follow-up interview at 2 months. Study participants will be contacted 2 months after their initial interview and provided with a follow-up survey that measures survival expectations, locus of control, and life satisfaction, mental health, savings, health behaviours, and (if applicable) schooling status. Participants will receive R50 in compensation for participation in the follow-up survey.

4. Surveillance Follow-up. Data from this study will be linked at the individual level to the AHRI population surveillance, which contains data on HIV testing, schooling, and employment. Participants will be visited approximately six weeks after the baseline survey and offered HIV testing as part of the AHRI surveillance. Passive follow-up through the surveillance is anticipated in future years, although this is beyond the scope of the registered trial. Linkage will be conducted by AHRI staff with access to identifying information in the population surveillance. After the conclusion of data collection and linkage, the key linking identifying data collected in this study to survey responses will be destroyed and only the de-identified ID number used in the demographic surveillance will remain. Participant contact details (not linked to data) will be retained in order to disseminate findings.

ELIGIBILITY:
Inclusion Criteria:

* resides in Africa Health Research Institute demographic surveillance area, specifically bounded structures to be visited during the last trimester of the surveillance in the "Southern PIPSA" area.
* member of a household in the AHRI demographic surveillance
* 18 to 25 years of age

Exclusion Criteria:

* <18, >25 years
* not a member of a household under surveillance
* not resident in the surveillance area

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 430 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bor, SD, Principal Investigator — Assistant Professor
Locations (1):
- Africa Health Research Institute, Somkhele, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be archived on the Africa Health Research Institute repository and will be available via a data request.
Supporting Information: Study Protocol
Time Frame: Data will be archived and publicly available within two years after data collection, and will be available indefinitely.
Access Criteria: Data use request to Africa Health Research Institute
URL: https://data.africacentre.ac.za

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from the population surveillance of the Africa Health Research Institute (AHRI) in Somkhele, South Africa, which served as the sampling frame.
Pre-assignment Details: From a pre-determined sample of 835 young adults, 433 young adults were found at home and a recruitment attempt was made. Of these, 430 consented to participate. 3 participants dropped out before completing the baseline survey, were not exposed to the treatment, and were blinded to their randomization status. 427 completed the baseline.
Period: Overall Study
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Started | 199 | 112 | 116
Completed | 199 | 112 | 116
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were either pre-populated (age, sex) based on information in the sampling frame or were collected via a baseline survey at time of enrollment into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control | Total
Number analyzed (Participants) | 199 | 112 | 116 | 427
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (2.1) | 21.1 (2.2) | 20.5 (2.1) | 20.8 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 63 | 62 | 229
  Male | 95 | 49 | 54 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Zulu-speaking, Black South African | 199 | 112 | 116 | 427
Region of Enrollment [Number; unit: participants]
  South Africa | 199 | 112 | 116 | 427
Subjective Life Expectancy at Baseline [Mean (Standard Deviation); unit: years] — Population: An error in the survey skip pattern led to substantial missing data in the first two weeks of data collection. This was identified during quality control checks, rectified, and enumerators were retrained. 27 of 35 missing values occurred in the first two weeks.
  years
    number analyzed (Participants) | 181 | 102 | 109 | 392
    (all) | 41.0 (12.0) | 40.0 (11.0) | 39.8 (12.0) | 40.4 (11.7)
Tested for HIV in Last 12 Months at Baseline [Count of Participants; unit: Participants] — Population: Totals differ due to item non-response.
  Participants
    number analyzed (Participants) | 198 | 111 | 115 | 424
    (all) | 116 | 64 | 77 | 257

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Participated in HIV Testing
Description: Participants were provided a voucher at baseline for free HIV testing at a private pharmacy in the area. This voucher could be used at any time within four weeks after baseline. Participants were also visited by an AHRI demographic and health surveillance team approximately six weeks after baseline during which all household members were offered a home-based rapid HIV test. This outcome takes the value of 1 if the participant used the HIV testing voucher OR participated in HIV testing during the household surveillance visit, and zero if the participant did not use the HIV testing voucher AND did not participate in HIV testing during the household surveillance visit.
Time Frame: 6 weeks
Population: All participants who completed the baseline survey, n=427.
Measure: Count of Participants; unit: Participants
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 199 | 112 | 116
Participants | 69 | 33 | 46

2. Secondary Outcome: Use of HIV Testing Voucher
Description: Participants were provided with a voucher for free HIV testing at a local service provider; use of voucher was assessed by obtaining voucher numbers and redemption dates from the service provider.
Time Frame: 4 weeks
Population: All participants completing the baseline survey, n=427.
Measure: Count of Participants; unit: Participants
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 199 | 112 | 116
Participants | 20 | 5 | 11

3. Secondary Outcome: Participation in HIV Testing or Care Services
Description: Same as primary outcome, but also including linkage to clinical HIV services (as assessed by the presence of a CD4 count)
Time Frame: 3 months
Population: Data were not collected.
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Attendance at Job Search Skills Workshop
Description: At the end of the baseline interview, participants were invited to a job search skills workshop facilitated by a local human resources consultant. Workshops were held at locations convenient to the study area and occurred 1-2 weeks after the baseline survey. Attendance was taken at the workshop. This outcome variable takes the value 1 if the participant attended the workshop and the value 0 if the participant did not attend the workshop.
Time Frame: 2 weeks
Population: All participants who completed the baseline survey, n=427.
Measure: Count of Participants; unit: Participants
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 199 | 112 | 116
Participants | 39 | 17 | 27

5. Secondary Outcome: Condoms Purchased
Description: At the end of the baseline survey, participants were offered the opportunity to purchase discount condoms. Participants were given 20 Rand and the opportunity to buy up to 10 condoms for 2 Rand each. The number purchased (0 to 10) was recorded.
Time Frame: Immediate post-test
Population: All participants who completed the baseline survey, n=427.
Measure: Mean (Standard Deviation); unit: condoms purchased
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 199 | 112 | 116
condoms purchased | 2.2 (2.7) | 2.3 (2.3) | 2.4 (2.7)

6. Secondary Outcome: Money Allocated to Savings Tin
Description: At the end of the baseline survey, participants were offered the opportunity to allocate a portion of their participation incentive (R100) to a savings tin. The amount saved was recorded. 13.5 Rands = 1 US dollar at the time of study.
Time Frame: Immediate post-test
Population: All participants who completed the baseline survey, n=427.
Measure: Mean (Standard Deviation); unit: Rand
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 199 | 112 | 116
Rand | 38.6 (29.1) | 43.1 (28.8) | 39.3 (29.4)

7. Secondary Outcome: Change in Subjective Life Expectancy (Baseline to Immediate Post-test)
Description: Subjective life expectancy was calculated as the under the subjective survival curve. Respondents were asked about the chances of surviving to age 30, 40, ..., 80 years. We linearly interpolated the responses and calculated the area under this curve, which we defined as subjective life expectancy (number of years expected to live between current age and age 80). Subjective life expectancy was elicited at baseline (pre-intervention), baseline (post-intervention), and at 8 weeks. This outcome measure reflects the immediate change in reported survival expectations induced by the intervention.
Time Frame: Baseline pre-test, Immediate post-test
Population: All participants who completed the baseline survey and had complete data for the survival expectations questions at baseline (pre-intervention) and immediate post-test, n=390.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 180 | 102 | 108
years | 1.3 (6.2) | 0.3 (6.4) | 0.7 (5.6)

8. Secondary Outcome: Subjective Life Expectancy (2 Months)
Description: Subjective life expectancy was calculated as the under the subjective survival curve. Respondents were asked about the chances of surviving to age 30, 40, ..., 80 years. We linearly interpolated the responses and calculated the area under this curve, which we defined as subjective life expectancy (number of years expected to live between current age and age 80). Subjective life expectancy was elicited at baseline (pre-intervention), baseline (post-intervention), and at 8 weeks. This outcome measure reflects the change in reported survival expectations at 8 weeks induced by the intervention.
Time Frame: 8 weeks
Population: Participants with non-missing survival expectations data in the baseline survey and 8-week follow-up survey, n=366.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
Number analyzed (Participants) | 167 | 95 | 104
years | -0.6 (11.8) | 0.6 (11.4) | 1.0 (11.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment through study completion at 8 weeks.
Description: Study staff reported adverse events through an anonymous reporting mechanism at AHRI. In addition, adverse events and protocol deviations were documented as part of daily field notes by the study team and reviewed by the study coordinator. Events were addressed when they occurred, and reported to the IRB when appropriate.
Arm/Group | A Beautiful Future Video | Active Control Video | Pure Control
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/112 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/112 | 0/116
Other Adverse Events (participants affected / at risk) | 0/199 | 0/112 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03215901/Prot_SAP_ICF_000.pdf